CLINICAL TRIAL: NCT03497065
Title: Awareness of Dental Implant Care and Its Correlation With Oral Hygiene Practices and the Presence of Peri-Implant Diseases
Brief Title: Dental Implant Care and Oral Hygiene Practices
Status: Completed | Type: Observational
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Jia Hui Fu, Associate Consultant, National University Health System, Singapore
Other Study IDs: 2017/00027
Record Dates: First submitted 2018-03-30; First posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Peri-implant Mucositis; Peri-Implantitis; Dental Plaque
Keywords: Dental devices; Home care; Awareness; Peri-implant mucositis; Peri-implantitis
MeSH Terms: conditions — Peri-Implantitis; Dental Plaque

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: non-surgical periodontal treatment — scaling, root planing, polishing, and oral hygiene education was performed

SUMMARY:
Objective: This study investigated how patients' knowledge, attitude, and perceptions influence their oral hygiene practices as well as peri-implant health. Materials and Methods: Participants with single implant crowns placed in 2007-2011 completed a questionnaire that examined their knowledge, attitude, and perceptions on oral hygiene practices and peri-implant health before receiving a periodontal examination, prophylaxis, and oral hygiene education. Clinical parameters recorded were peri-implant probing depths and plaque index, width of keratinized mucosa, implant crown characteristics, reason for tooth loss, and diagnosis of peri-implant health.

DETAILED DESCRIPTION:
First, a trained clinical research dental assistant interviewed the participants and showed them pictures of oral hygiene aids so that the participants could answer the survey questions accurately. Subsequently, a periodontal examination, dental prophylaxis, and oral hygiene education were performed. Participants with active diseases e.g. caries, periodontitis, or peri-implantitis were referred for further management. The following clinical parameters were recorded during the examination:

1. Probing depths at 6 sites around the implant (mesiobuccal, midbuccal, distobuccal, distolingual, midlingual and mesiolingual)
2. Plaque index (Silness & Loe 1964) at 4 sites around the implant (mesial, buccal, distal and lingual)
3. Amount of keratinized mucosa at the implant site
4. Characteristics of the implant crown:

   * Type of implant crown (screw- or cement-retained) and
   * Position of crown margins (supra-, equi- or sub-gingival)
5. Reason(s) for tooth loss
6. Diagnosis of peri-implant health

   * Normal
   * Mucositis, defined as 3 or more bleeding points per implant
   * Peri-implantitis, defined as implant thread exposure that was either clinically visible or detectable with a periodontal probe.

ELIGIBILITY:
Inclusion Criteria:

* English speaking patient
* Aged 21 years old or above
* Received at least 1 implant-supported single crown from NUH in the year 2007-2011 (in functional loading for at least 5 years)

Exclusion Criteria:

* Implant is used to restore overdentures or multi-unit restorations such as splinted crowns, fixed partial dentures, and cantilevers.
* Pregnant/lactating women
* Parkinson's disease or any other debilitating diseases
* Physical or mental disabilities that may impair oral hygiene practices
* Poorly controlled diabetes
* Heavy smoker (10 or more cigarettes per day)
* Radiation therapy in head and neck region
* HIV, TB, hepatitis or other infectious diseases
* Drug and alcohol abuse

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population is made up 50.6% male and 49.4% female, mainly Chinese (87.3%), Indian (5%), Malay (3.8%), Caucasian (1.3%), Eurasian (1.3%), and Japanese (1.3%), with a mean age of 58.6 years old.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
qualitative assessment of patient's knowledge on care and maintenance of dental implants using a questionnaire based on a 5 point Likert scale | 1 day
  patient's knowledge of peri-implant diseases

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No